CLINICAL TRIAL: NCT02434562
Title: Development and Validation of in Vitro Cell-based Bioassays for Nuclear Receptor Activation by Human Serum
Brief Title: Development and Validation of in Vitro Cell-based Bioassays for Nuclear Receptor Activation
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s54034
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2016-05

CONDITIONS: Hypogonadism; Estrogens; Testosterone; Androgens
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Medical castration: Patients treated with androgen deprivation therapy (e.g. for hypersexuality, transgender subjects, ...)
  Interventions: Other: Serum (with or without urine) samples
- Male hypogonadism: Patients treated with testosterone replacement therapy (e.g. for late-onset hypogonadism, secondary hypogonadism)
  Interventions: Other: Serum (with or without urine) samples
- Thyroid disorders: Patients treated for hyperthyroidism or hypothyroidism (incl. during treatment for thyroid cancer)
  Interventions: Other: Serum (with or without urine) samples
- Obesity and weight loss: Patients treated for obesity with weight loss interventions (mainly bariatric surgery)
  Interventions: Other: Serum (with or without urine) samples
- Miscellaneous: Various disorders associated with alterations in SHBG, androgens and/or estrogens

INTERVENTIONS:
Other: Serum (with or without urine) samples
  Groups: Male hypogonadism; Medical castration; Obesity and weight loss; Thyroid disorders

SUMMARY:
This is a prospective biobank set up to collect serum from patients with disorders associated with changes in androgens, estrogens or sex hormone-binding globulin (SHBG), before and/or after treatment.

DETAILED DESCRIPTION:
In vitro cell-based bioassays may be a technique to measure serum androgen or estrogen bioactivity. In this study investigators are collecting serum (and if possible, urine) samples from different cohorts of patients, before and/or after treatment.

The aim is to measure androgens, estrogens and SHBG as well as in vitro bioactivity with newly developed cell-based bioassays, and to compare different techniques to each other as well as to clinical endpoints available in the patient's Electronic Health Record.

ELIGIBILITY:
Inclusion Criteria:

* Known or expected medical condition affecting androgens, estrogens or SHBG

Exclusion Criteria:

* Inability to provide written informed consent
* Known or suspected bloodborne infectious diseases (e.g. HIV, viral hepatitis etc.)
* Anemia (<11 g/dL hemoglobin) or being a Jehovah's Witness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the department of Endocrinology/Andrology, Urology and Oncology
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2012-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Testosterone bioequivalents (in nanomolar) | second blood sample at time of clinical follow-up (between 3 weeks and 1 year interval)
Estradiol bioequivalents (in picomolar) | second blood sample at time of clinical follow-up (between 3 weeks and 1 year interval)

SECONDARY OUTCOMES:
Calculated free and bioavailable testosterone (in nanomolar) | second blood sample at time of clinical follow-up (between 3 weeks and 1 year interval)
Calculated free and bioavailable estradiol (in picomolar) | second blood sample at time of clinical follow-up (between 3 weeks and 1 year interval)
Total serum testosterone (in nanomolar) | second blood sample at time of clinical follow-up (between 3 weeks and 1 year interval)
  Measured by immunoassay or liquid chromatography tandem mass spectrometry (LC-MS/MS)
Total serum estradiol (in picomolar) | second blood sample at time of clinical follow-up (between 3 weeks and 1 year interval)
  Measured by immunoassay or LC-MS/MS
Total serum SHBG (in nanomolar) | second blood sample at time of clinical follow-up (between 3 weeks and 1 year interval)
  Measured by immunoassay

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Vanderschueren, MD, PhD, Principal Investigator — UZ Leuven

REFERENCES:
- [Result] Laurent MR, Helsen C, Antonio L, Schollaert D, Joniau S, Vos MJ, Decallonne B, Hammond GL, Vanderschueren D, Claessens F. Effects of sex hormone-binding globulin (SHBG) on androgen bioactivity in vitro. Mol Cell Endocrinol. 2016 Dec 5;437:280-291. doi: 10.1016/j.mce.2016.08.041. Epub 2016 Aug 26. PMID 27576188